CLINICAL TRIAL: NCT03871010
Title: Midline Programme - Vascular Nursing Team
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: KHO-02-Midline; RVO-FNOs/2017 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Inflammation; Local; Infection
Keywords: Midline catheter; Vascular nursing team
MeSH Terms: conditions — Inflammation; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neutropenia patients, Dept. of Haematooncology: Patients with neutropenia from the Department of Haematooncology were included in this group.
  Interventions: Device: Midline catheter
- No neutropenia patients, Dept. of Haematooncology: Patients without neutropenia from the Department of Haematooncology were included in this group.
  Interventions: Device: Midline catheter
- No neutropenia patients, other clinical depts.: Patients with neutropenia from the other clinical departments of the University Hospital Ostrava were included in this group.
  Interventions: Device: Midline catheter

INTERVENTIONS:
Device: Midline catheter — Midline catheter is used for administration of intravenous therapy, and is inserted in a larger vein.

SUMMARY:
Integration of the Vascular Nursing Team of the Department of Haematooncology, University Hospital Ostrava for the needs of all clinical departments of the hospital. Assessment of local signs of inflammation in patients of the Department of Haematooncology and other clinical departments of the University Hospital Ostrava.

DETAILED DESCRIPTION:
The study subjects were indicated by a physician for Midline catheter insertion.

Prior to insertion of the catheter, the study subjects were fully informed and signed the informed consent with participation in the study.

Local signs of inflammation were recorded in the study subjects, together with basic demographic characteristics (age, sex, diagnosis), and complications during catheter insertion, the number of days when the Midline catheter was inserted, number of changes of the dressings, presence of neutropenia in the study subjects and the score of local inflammation according to Madonna.

* Degree 0- no pain or reaction in the surrounding
* Degree 1 - pain only, no reaction in the surrounding
* Degree 2 - pain and reddening
* Degree 3 - pain, reddening, swelling or painful stripe along the vein
* Degree 4 - puss, swelling, reddening and painful stripe along the vein The investigators also observed on which day the first signs of infection appeared.

ELIGIBILITY:
Inclusion Criteria:

* insertion of Midline catheter by nurses from the Vascular Nursing Team
* age over 18 years

Exclusion Criteria:

- inability to insert the Midline catheter

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Midline catheter hospitalized at clinical department of the University Hospital Ostrava, Czech Republic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Local signs of infection | 3 days at minimum
  Local signs of infection were recorded, using the scoring system according to Madonna - see detailed description.

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Hašová, Mgr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to make individual participant data available to other researchers.